CLINICAL TRIAL: NCT05095168
Title: Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of a Single Ascending Dose (SAD) of CAN106 Administered Intravenously (IV) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CARE Pharma Shanghai Ltd. (Industry)
Responsible Party: Sponsor
Organization: CANbridge Life Sciences Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN106-HV-101
Record Dates: First submitted 2021-09-22; First posted 2021-10-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: PNH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): In the SAD arm subjects will be sequentially included in one of up to six cohorts (dose levels). Additional subjects may be added in any cohort if necessary.
  Interventions: Drug: CAN106
- placebo (Placebo Comparator): In the SAD arm subjects will be sequentially included in one of up to six cohorts (dose levels). In higher dose levels, subjects will be randomized to receive the treatment or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAN106 — CAN106 is a selective inhibitor of complement activation, which binds to the complement component C5.
  Arms: Single Ascending Dose (SAD)
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
This is a single site, single dose escalation study in healthy subject with CAN106. The study is to assess the safety and tolerability of single escalating doses of CAN106; to characterize the PK and PD profile of CAN106; and to evaluate the immunogenicity of CAN106 injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and provide informed consent.
* Males or females, between 21 and 45 years of age, inclusive;
* Body mass index must be within the range of 18.5 to 32.0 kg/m2;
* 12-lead electrocardiogram (ECG) within normal limits with no clinically significant abnormalities in the opinion of the Investigator；
* Systolic blood pressure ≤140 mmHg and a diastolic blood pressure of ≤ 90 mmHg after 5 minutes with supine rest；
* non-pregnancy
* meningococcal vaccinations for at least 2 weeks before dosing

Exclusion Criteria:

* Disease or conditions interfere with participating the trial
* Active serious mental illness or psychiatric disorder
* clinically relevant abnormal test results in hepatic function
* unacceptable CBC lab test
* asymptomatic complement deficiency
* Any other clinical safety laboratory test
* HIV, HBV, HCV positive
* Alcohol and drug abuse
* etc.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects with dose-limiting toxicity (DLTs) | 6-months after dosing
  TEAEs will be categorized as per the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria.
  a DLT is defined as one subject with a Grade 3 AE or higher, that are assessed as drug-related by the site investigator.
Incidence of adverse events (AEs) | 6-months after dosing
  An AE is defined as any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Incidence of severe adverse events (SAEs) | 6-months after dosing
  Any untoward medical occurrence that at any dose:
  * Results in death,
  * Is life-threatening,
  * Requires inpatient hospitalization or prolongation of existing hospitalization,
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect. (ICH E6 (R2))

SECONDARY OUTCOMES:
PK parameters - tmax | 6-months after dosing
  time to reach maximum of concentration (days)
PK parameters-Cmax | 6-months after dosing
  peak plasma concentration
PK parameters - AUC0-t | 6-months after dosing
  Area under the plasma concentration versus time curve to the last visit (AUCt)
PK parameters - t1/2 | 6-months after dosing
  terminal elimination half-life
PD endpoints-free C5 | 6-months after dosing
  maximal change from baseline in free C5 concentrations at each of scheduled post baseline assessment time-points (µg/ml);
PD endpoints-CH50 | 6-months after dosing
  maximal change from baseline total complement activity (CH50) at each of scheduled post baseline assessment time-points (%);
PD endpoints-total C5 | 6-months after dosing
  meausure the absolute change from baseline in total C5 concentrations at each of scheduled post baseline assessment time-points (µg/ml);
Immunogenicity | 6-months after dosing
  Anti-drug Antibody (ADA) titers

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore